CLINICAL TRIAL: NCT00827034
Title: A Phase 1, Randomized, Open-Label, Two-Way Crossover Study To Evaluate The Steady-State Effect Of Dimebon (PF 01913539) On The Single-Dose Pharmacokinetics And Pharmacodynamics Of Warfarin In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B1451020
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer's Disease; Huntington's Disease
Keywords: Dimebon Warfarin Drug-Drug Interaction
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease | interventions — Warfarin; latrepirdine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): A: Warfarin alone
  Interventions: Drug: Warfarin
- B (Other): B: Dimebon and Warfarin co-administration
  Interventions: Drug: Dimebon; Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — A: a single oral dose of warfarin 25 mg administered on Day 1 of the relevant dosing period, as tablets.
  Arms: A
Drug: Dimebon — B is oral doses of Dimebon 10 mg TID on Days 1 7 and Dimebon 20 mg TID on Days 8 17, with co administration of a single oral dose of warfarin 25 mg on Day 12 of the relevant dosing period, both as tablets
  Arms: B
Drug: Warfarin — B is oral doses of Dimebon 10 mg TID on Days 1 7 and Dimebon 20 mg TID on Days 8 17, with co administration of a single oral dose of warfarin 25 mg on Day 12 of the relevant dosing period, both as tablets
  Arms: B

SUMMARY:
This study will evaluate the potential drug-drug interaction of Dimebon with the FDA-recommended CYP2C9 substrate warfarin in healthy subjects. Conformance with the guidance includes general study design using a randomized, open label, single-dose warfarin, steady-state Dimebon, 2-sequence, 2-treatment, 2-period crossover design with a minimum 7-day washout period between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Prothrombin time (PT)/INR, and partial thromboplastin time (PTT).
* Plasma Protein C and Protein S activity (functional) within the normal reference range.

Exclusion Criteria:

* A known sensitivity or previous intolerance to Dimebon or warfarin.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Subjects receiving warfarin for treatment of active thromboembolic events (ie, pulmonary embolism, deep vein thrombosis), as well as subjects anticoagulated with prosthetic heart valves.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Single dose pharmacokinetics (Cmax, AUCinf) of warfarin 25 mg with and without co-administration of steady-state Dimebon 20 mg TID in healthy adult subjects. | 7+18 days
Single dose pharmacodynamics (INRmax, AUC-INR) of warfarin 25 mg with and without co-administration of steady-state Dimebon 20 mg TID in healthy adult subjects. | 7+18 days
Safety and tolerability ( adverse event monitoring, physical examinations, vital signs, ECG's and clinical laboratory tests) of multiple doses of Dimebon 20 mg TID with a single dose of warfarin 25 mg in healthy adult subjects. | 7+18 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451020